CLINICAL TRIAL: NCT06651684
Title: A Randomized Controlled Trial of a Smoking Cessation Intervention Including Health Navigators to Address Unmet Social Needs of Parents Who Smoke
Brief Title: Smoking Cessation Intervention Including Health Navigators to Address Unmet Social Needs of Parents Who Smoke
Acronym: CanCEASE-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Olivier Drouin, M.D., M.Sc M.P.H., Pediatrician and Clinical Assistant Professor, Departments of Paediatrics and Department of Social and Preventive Medicine, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MP-21-2025-7715; 506937 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-10-04; First posted 2024-10-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Smoking Cessation; Tobacco Dependence
Keywords: Smoking cessation; Social risk; Second hand smoke; Health navigator; Unmet social needs
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Pragmatic, single-blind
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Care-as-usual (No Intervention): Participants assigned to this group will receive care as usually delivered in participating clinics and list of smoking cessation resources, including instructions to access Nicotine Replacement Therapy (NRT).
- CanCEASE with Health Navigator (Experimental): Participants assigned to this arm will receive smoking cessation resources, including instructions to access Nicotine Replacement Therapy (NRT) at Baseline, 6 and 12 months. They will also have the choice to schedule support sessions with a Health Navigator, which will be an individual with lived experience related to tobacco and trained to provide support for unmet social needs.
  Interventions: Behavioral: CanCEASE with Health Navigator

INTERVENTIONS:
Behavioral: CanCEASE with Health Navigator — CanCEASE is a digital intervention to identify parents who smoke, assess their motivation and willingness to quit, as well as to provide direct linkage to evidence-based smoking interventions, including effective behavioural and pharmacological resources that can be used alone or in combination.
  Participants will have the choice to receive CanCEASE at three timepoints (0, 6 and 12 months). CanCEASE will be combined with an offer of support sessions with a Health Navigator.
  Health Navigators will be research personnel hired specifically for this study and trained formally in health navigation, tobacco cessation counseling and strategies to address unmet social needs. The investigators will leverage knowledge and experience of two ongoing RCTs of HNs in pediatrics to inform training strategies.
  Arms: CanCEASE with Health Navigator

SUMMARY:
Background: The goal of this study is to address parental smoking and social adversity, which can present an obstacle for smoking cessation, in order to decrease childhood exposure to second-hand cigarette smoke. To address these factors, this study includes a smoking cessation intervention for parents and legal guardians recruited in pediatric clinics (CanCEASE), as well as the support of a Health Navigator (HN) to work with the participant towards the resolution or mitigation of unmet social needs.

Participants: The research team will recruit one thousand participants from pediatric outpatient clinics within two healthcare centres in and around the city of Montreal, Canada, over the course of 2.5 years. Eligible persons are parents and legal guardians, of any sex and gender, accompanying children under 18 to their scheduled medical appointments, and who report at least one social risk in selected areas (i.e., employment, housing stability, ability to pay for utilities, financial resource strain, food security, transportation, childcare, parent education and health literacy). Participants must also be 18 years old or older with sufficient proficiency in French or English to complete the interviews and questionnaires. In households in which both parents smoke, only one will be eligible to participate, but smoking cessation information will be offered to both. Families presenting at the clinic for an urgent medical issue are not eligible to participate.

Intervention: Participants will be divided into control group (care as usual with CanCEASE at the end of the study period) and intervention (CanCEASE + Health navigator). All participants will complete questionnaires at Baseline, 6 and 12 months. The intervention group will receive CanCEASE at the end of each questionnaire. Controls will receive CanCEASE at 12 months. The intervention group will have the possibility to meet with the HNs and will be invited to commit to at least two sessions (i.e.: evaluation and a follow up), with the option to book more time as needed.

Aims and hypotheses: Examining how effective the combination of CanCEASE with HN support is in helping parents with unmet social needs quit smoking. Investigators will also examine the effects of the intervention on status of unmet social needs, if the intervention was implemented as planned and well accepted by clinics and participants, and what is the cost of the intervention for each person who quits smoking.

DETAILED DESCRIPTION:
Primary purpose: The overarching goal of the study is to address child second-hand-smoke exposure by supporting parent smoking cessation. For that purpose, the investigators designed the present investigator-blinded, randomized controlled clinical trial, to be carried out in real-world settings, in order to test the effectiveness of two combined interventions, one to promote smoking cessation and another to support parents with unmet social needs, which could be hindering their smoking cessation efforts.

Rationale: In Canada, tobacco use is the greatest cause of preventable morbidity and mortality, generating attributable annual health-related costs of CAD $16.2 billion and 48 thousand deaths. Parental smoking has direct impacts on child health, starting at in-utero stages (e.g., fetal growth restriction, premature birth, sudden infant death syndrome, and exacerbation of respiratory illnesses) and it contributes to child and adolescent smoking initiation. Yet, despite its well-known negative effects, 15% of Canadian children are exposed to household second-hand smoke. Data also indicate that parents are overall underserved in terms of medical care and see their child(ren)'s medical care providers more often than their own, but they are not frequently screened for smoking (less than 5% of visits to pediatric practices) nor do they receive any smoking cessation support. Yet, twenty-five percent of all adult smokers have children who are seen in child healthcare offices. Further, smoking and social economic status (SES) are strongly associated, such that populations with lower SES present higher proportions of tobacco use, indicating lower SES can be an obstacle to smoking cessation as well as a perpetuating factor for smoking.

Aims and hypotheses:

Aim 1 - Examining the effectiveness of the intervention (CanCEASE + HN) on smoking cessation compared to care-as-usual. Hypothesis 1: the intervention will lead to a higher proportion of quits among smoking parents than the control condition.

Aim 2 - Examining the effectiveness of the intervention (HN) on unmet social needs and, if so, does the resolution of an unmet social need mediate CanCEASE-related smoking cessation. Hypotheses: (2a) there will be a greater decrease in the prevalence of unmet social needs in the intervention vs. control arm; (2b) resolution of unmet social need(s) will mediate in part the effect of the intervention on smoking cessation.

Aim 3 - Assessing whether the intervention (CanCEASE + HN) implemented as planned is acceptable to participants and practices. Hypotheses: (3a) both intervention and control will be acceptable to participants and practices where they are implemented; (3b) both the intervention and control will be delivered as planned to most participants.

Aim 4 - Examining the incremental cost-effectiveness ratio in Canadian dollars per quit of CanCEASE with HN compared to care-as-usual. Hypothesis 4: The intervention will have a favorable cost per quit compared to control.

Participant recruitment: Participants (N=1000) will be recruited from pediatric outpatient clinics in two healthcare centres in Montreal, Canada (i.e., General pediatrics outpatient clinic, CHU Sainte-Justine; Outpatient pediatric clinics, Hôpital Maisonneuve-Rosemont). Potential participants will initially undergo a brief pre-screening process that should take under a minute to complete. It is designed for initial identification of parents who smoke using questions about data on relationship of the child with the accompanying adult, smoking status of the adult and contact information. This first pass prevents adults in the clinic from spending too much time in activities unrelated to their visit and prevents disruption of the work flow at the recruiting sites. Pre-screening can be completed via the study website, self-check-in stations in the recruitment sites (where available), and via the hospital appointment confirmation systems. Alternatively, pre-screening will be conducted by an on-site research assistant when parents come to register for an appointment. Recruitment will also be done via referral by the clinical or front desk teams either by having interested individuals fill out an "authorization to contact form" or by scanning a QR code from posters that will be placed in the clinics, such that the research team can contact potential participants to present the study, obtain informed consent, assess them for social risks to determine if the individual is eligible to participate in the study.

Intervention: CanCEASE is a parental smoking cessation intervention that facilitates referral and linkage to existing healthcare and community resources and it is available in both French and English. It consists of (1) asking about smoking status, (2) a self-assessment of readiness to quit, and interest in available resources, (3) providing advice on available services with brief motivational messages, (4) assistance to quit, via quit lines and text message support, and (5) assistance with access to Nicotine Replacement Therapy (NRT). Participants will be randomized either to the control or the intervention arm of the study. In both arms, participants will complete three questionnaires, one within the first month after recruitment, then 6 and 12 months later. CanCEASE will be offered after the end of each questionnaire to participants in the intervention arm of the study and after the 12-month questionnaire to control participants. Control group will receive care-as-usual, depending on what is typically available on site, and at recruitment, a resource list with freely available cessation resources with advice on how to obtain NRT. Participants in the intervention group will receive, in addition to CanCEASE, two support sessions a health navigator (HN). HNs are individuals trained in specific areas of health, but who do not necessarily hold a professional degree. Their role is to provide assistance in ways that are complementary to what an individual receives from the healthcare system. HNs can potentially enhance smoking cessation efforts by facilitating access to resources and supporting participants facing poverty-related challenges that hinder their cessation efforts. Participants are expected to commit to at least two sessions with the HN, the initial evaluation and follow up. Session 1 will take place about 14 days after baseline questionnaire, according to participant availability. It will consist of an evaluation, information session, specification of quitting goals and specifying unmet social needs. During and, if needed, on the days following the session, the HN will facilitate participant access to resources and send support materials as needed. Session 2 will occur about a month after baseline questionnaire, according to participant availability. At this time, the HN will go over the current smoking and unmet needs status, inquire about barriers and challenges, and will follow-up on referrals and resources that were previously provided. Participants are free to book additional HN sessions as needed for as long as they are actively taking part in the study. After every session, participants will receive a satisfaction survey to fill out. Whenever a participant reports having quit smoking, they will be invited to provide a urine sample for lab confirmation that there is no longer any nicotine in their system. Urine samples will be self-collected and sent by accelerated postage.

Relevance: This RCT will compare, in families with unmet social needs, the effectiveness and cost-effectiveness of the CanCEASE intervention for parental smoking cessation with HN support in comparison to care as usual plus information on freely available cessation resources. It could yield data that supports leveraging implementation of preventive primary care to improve population health.

ELIGIBILITY:
Inclusion Criteria:

* Parents or legal guardians aged ≥18 years, with child(ren) aged 0-17 years, attending a regular scheduled medical appointment in one of the study sites.
* Smokers with at least one self-reported social risk as assessed by validated screening questions on the domains employment, housing stability, ability to pay for utilities, financial resource strain, food security, transportation, childcare, parent education and health literacy.
* Sufficiently proficient in French or English to understand and complete study questionnaires.

Exclusion Criteria:

* Families presenting at the clinic for an urgent medical issue.
* Parents without at least one social risk.
* If both parents smoke, only one parent will be eligible to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Aim 1 - 7-day abstinence | 6 months; 12 months
  Percentage of participants who self-report 7-day abstinence
Aim 1 - Smoking intensity | 0 months; 6 months; 12 months
  Average self-reported number of cigarettes per day.
Aim 1 - Cotinine-confirmed quit | 6 months; 12 months
  Urinary cotinine values below 100 ng/ml, a consensus cutoff level, biochemical confirmation of 7-day abstinence.
Aim 1 - Anabasine-confirmed quit | 6 months; 12 months
  Urinary anabasine detection allows for the differentiation between smokers and abstainers who are using NRT at concentrations below 1.2 ng/mL.
Aim 1 - Quit attempts | 6 months; 12 months
  Percentage of participants who report at least one 24-hour quit.
Aim 1 - Intent to quit | 0 months; 6 months; 12 months
  Percentage of parental smokers who are seriously considering quitting in the next six months.
Aim 2 - Resolution of social risk | 12 months
  Percentage of participants who report resolution of one or more social risks at the end of the study. Outcome will be calculated via the comparison of Social Risk questionnaire responses at baseline and at 12 months to determine persistence of social risk (no longer reported=yes; still reported=no).
Aim 2 - Improvement in unmet social needs | 12 months
  Self-reported improvement in unmet social need present at baseline on a 5-point Likert scale wherein: 1=Much better, 2=Somewhat better, 3=Stayed the same, 4=Somewhat worse, 5=Much worse.
Aim 2 - Access to resources to help with unmet social needs | 12 months
  Percentage of participants who, at follow-up, self-report having accessed 1+ resources for each unmet social needs present at baseline
Aim 3 - Interest in resources to help them quit | 0 months; 6 months; 12 months
  Percentage of participants who are interested in referral to quitline or text-message cessation program (SMAT) and/or prescription of pharmacotherapy to help quit (NRT)
Aim 3 - Meaningful receipt of assistance | 6 months; 12 months
  Percentage of participants who, at follow-up, self-report having received at least one of the following: referral to quitline or text-message cessation program (SMAT) or prescription of pharmacotherapy to help quit (NRT).
Aim 3 - Proportion or participants who had contact with HNs | 12 months
  Percentage of participants who, at follow-up, self-report having received at least one session with health navigator (Intervention arm only)
Aim 3 - Number of sessions with heath navigators | 12 months
  For each participant, number of sessions with the health navigator (Intervention arm only).
Aim 3 - Duration of sessions with heath navigators (in minutes) | 12 months
  For each participant, the average number of minutes per session health navigators spent with participants on average (Intervention arm only).
Aim 4 - Incremental cost-effectiveness ratio - intervention vs. usual care (from a healthcare system perspective) | Through study completion, an average of 1 year
  Difference in costs (intervention minus control) divided by difference in effectiveness (intervention minus control). Reported in Canadian dollars per quit.
  Costs will include both material and personnel costs. Personnel costs will be obtained by multiplying the total time devoted to interventions/usual care activities by national average wage rate for each type of personnel.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Drouin, MD, MSc, MPH, Principal Investigator — CHU Sainte-Justine Research Centre; Nicholas Chadi, MD, MPH, Principal Investigator — CHU Sainte-Justine Research Centre
Locations (2):
- Canada (2):
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Pediatric Clinic of the CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No